CLINICAL TRIAL: NCT04337229
Title: Evaluation of Comfort Behavior Levels of Newborns With Artificial Intelligence Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, DENİZ YİĞİT, Research Assistant, Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DYIGIT; Ayfer ACIKGOZ (Other: Eskişehir Osmangazi Üniversitesi)
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Newborn; Comfort; Nursing; Artificial Intelligence
Keywords: newborn; comfort; nursing; artificial intelligence

STUDY DESIGN:
Intervention Model Description: it is planned to create a technology that determines the comfort level of the newborn quickly and simply, easy to use, time-saving and can be used by the mobile device.
Masking Description: Researchers and family of newborns will know about all the details of the study. Verbal and written permission will be obtained from families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- artificial intelligence techniques (Experimental): Facial and body movements of newborns will be recorded by camera, and images will be processed in computer environment by using artificial intelligence techniques. As a result, it is planned to create a technology that determines the comfort level of the newborn quickly and simply and can be used by the mobile device.
  Interventions: Other: Artifical intelligent

INTERVENTIONS:
Other: Artifical intelligent — it is planned to create a technology that determines the comfort level of the newborn quickly and simply, easy to use, time-saving and can be used by the mobile device.

SUMMARY:
This study; It will be carried out with the aim of developing the artificial intelligence method, which allows automatic determination of comfort levels of newborns.

DETAILED DESCRIPTION:
This study; It will be carried out with the aim of developing the artificial intelligence method, which allows automatic determination of comfort levels of newborns. Facial and body movements of newborns will be recorded by camera, and images will be processed in computer environment by using artificial intelligence techniques. As a result, it is planned to create a technology that determines the comfort level of the newborn quickly and simply and can be used by the mobile device.

ELIGIBILITY:
Inclusion Criteria:

* Parents' acceptance of their baby's participation in the study
* Having a baby born at 24-42 weeks

Exclusion Criteria:

* Having a baby born before 24 weeks of gestation or after 42 weeks of gestation.
* Has received analgesic, muscle relaxant or sedative drug treatment that may affect comfort and behavior (last 24 hours)
* Newborn has serious neurological damage

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Images of the newborn | 12 hours for each newborn
  Images will be taken to transfer behaviors of newborns to the computer. Attention will be paid to making face and body movements visible while taking the image.The camera will take 12 hours of view of each newborn.However, this period can be shortened as a result of preliminary work.

SECONDARY OUTCOMES:
Artificial intelligence techniques | Approximately 1 week for each newborn
  The images of the newborn will be transferred to the computer. The images will be processed by a specialist on computer using artificial intelligence techniques.

CONTACTS AND LOCATIONS:
Overall Officials: DENİZ YİĞİT, Res.Asst., Principal Investigator — ESKİŞEHİR OSMANGAZİ ÜNİVERSİTESİ SAĞLIK BİLİMLERİ FAKÜLTESİ

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, it is aimed to announce the artificial intelligence developed to measure comfort with the declaration to be made in international congresses. In this way, it is thought that the program will be used by healthcare professionals in different hospitals and neonatal clinics in these hospitals.
Supporting Information: Study Protocol
Time Frame: It will be shared after the study is finished (About 2 years later)
Access Criteria: Being a healthcare professional working with newborns

REFERENCES:
- [Result] Ambuel B, Hamlett KW, Marx CM, Blumer JL. Assessing distress in pediatric intensive care environments: the COMFORT scale. J Pediatr Psychol. 1992 Feb;17(1):95-109. doi: 10.1093/jpepsy/17.1.95. PMID 1545324
- [Result] Arroyo-Novoa CM, Figueroa-Ramos MI, Puntillo KA, Stanik-Hutt J, Thompson CL, White C, Wild LR. Pain related to tracheal suctioning in awake acutely and critically ill adults: a descriptive study. Intensive Crit Care Nurs. 2008 Feb;24(1):20-7. doi: 10.1016/j.iccn.2007.05.002. Epub 2007 Aug 6. PMID 17689249
- [Result] Arslan, H., & Konuk Şener, D. (2009). Stigma, spiritüalite ve konfor kavramlarının Meleis' in kavram geliştirme sürecine göre irdelenmesi. Maltepe Üniversitesi Hemşirelik Bilim ve Sanatı Dergisi, 2(1): 51-58.
- [Result] Atalay, M., & Çelik, E. (2017). Büyük veri analizinde yapay zekâ ve makine öğrenmesi uygulamaları. Mehmet Akif Ersoy Üniversitesi Sosyal Bilimler Enstitüsü Dergisi, 9(22): 155-172.
- [Result] Aydın, Ş.E. (2017). Yapay zeka teknolojisi (yapay zekaların dünü bugünü yarını), Yüksek lisans tezi, Çukurova Üniversitesi, Adana.
- [Result] Bodur, G., & Kaya, H. (2017). Hemşirelerin gözüyle gelecek: 2050'li yıllar. Ege Üniversitesi Hemşirelik Fakültesi Dergisi, 33 (1): 27-38.
- [Result] Coughlin M, Gibbins S, Hoath S. Core measures for developmentally supportive care in neonatal intensive care units: theory, precedence and practice. J Adv Nurs. 2009 Oct;65(10):2239-48. doi: 10.1111/j.1365-2648.2009.05052.x. PMID 19686402
- [Result] Çınar Yücel Ş. (2011). Kolcaba'nın konfor kuramı. Ege Üniversitesi Hemşirelik Yüksek Okulu Dergisi, 27: 79-88.
- [Result] Çimen, Ü. (2016). Solunum seslerinin yapay zekâ ortamında sınıflandırılması, Yüksek Lisans Tezi, Afyon Kocatepe Üniversitesi Fen Bilimleri Enstitüsü, Afyonkarahisar.
- [Result] de Sousa Freire NB, Garcia JBS, Lamy ZC. Evaluation of analgesic effect of skin-to-skin contact compared to oral glucose in preterm neonates. Pain. 2008 Sep 30;139(1):28-33. doi: 10.1016/j.pain.2008.02.031. Epub 2008 Apr 22. PMID 18434021
- [Result] Hunter, J. (2010). Therapeutic positioning: neuromotor, physiologic, and sleep implications. Developmental care of newborns and infants. A guide for health professionals. 2nd edn. Glenview, IL: NANN: 283-312.
- [Result] Ista E, van Dijk M, Tibboel D, de Hoog M. Assessment of sedation levels in pediatric intensive care patients can be improved by using the COMFORT "behavior" scale. Pediatr Crit Care Med. 2005 Jan;6(1):58-63. doi: 10.1097/01.PCC.0000149318.40279.1A. PMID 15636661
- [Result] Kahraman, A., Başbakkal, Z., & Yalaz, M. (2014). Yenidoğan konfor davranış ölçeği'nin Türkçe geçerlik ve güvenirliği. Uluslararası Hakemli Hemşirelik Araştırmaları Dergisi, 1(2).
- [Result] Karabacak, Ü., & Acaroğlu, R. (2011). Konfor kuramı. Maltepe Üniversitesi Bilim ve Sanat Dergisi, 4(1): 197-202.
- [Result] Karakaplan, S., & Yıldız, H. (2010). Doğum sonu konfor ölçeği geliştirme çalışması. Maltepe Üniversitesi Hemşirelik Bilim ve Sanatı Dergisi, 3(1): 55-65.
- [Result] Kaya, U., Yılmaz, A., & Dikmen, Y. (2019). Sağlık alanında kullanılan derin öğrenme yöntemleri. Avrupa Bilim ve Teknoloji Dergisi, (16): 792-808.
- [Result] Kolcaba K, DiMarco MA. Comfort Theory and its application to pediatric nursing. Pediatr Nurs. 2005 May-Jun;31(3):187-94. PMID 16060582
- [Result] Kolcaba K, Tilton C, Drouin C. Comfort Theory: a unifying framework to enhance the practice environment. J Nurs Adm. 2006 Nov;36(11):538-44. doi: 10.1097/00005110-200611000-00010. PMID 17099440
- [Result] Kuğuoğlu, S., & Karabacak, Ü. (2008). Genel konfor ölçeğinin Türkçe'ye uyarlanması. İ.Ü.F.N. Hemşirelik Dergisi, 16 (61): 16-23.
- [Result] Küçük Alemdar, D., & Güdücü Tüfekçi, F. (2015). Prematüre bebek konfor ölçeği'nin Türkçe geçerlilik ve güvenilirliği. Hemşirelikte Eğitim ve Araştırma Dergisi, 12 (2): 142-148.
- [Result] Losacco V, Cuttini M, Greisen G, Haumont D, Pallas-Alonso CR, Pierrat V, Warren I, Smit BJ, Westrup B, Sizun J; ESF Network. Heel blood sampling in European neonatal intensive care units: compliance with pain management guidelines. Arch Dis Child Fetal Neonatal Ed. 2011 Jan;96(1):F65-8. doi: 10.1136/adc.2010.186429. PMID 21177753
- [Result] Mathai S, Natrajan N, Rajalakshmi NR. A comparative study of nonpharmacological methods to reduce pain in neonates. Indian Pediatr. 2006 Dec;43(12):1070-5. PMID 17202604
- [Result] Mijwel, M. M. (2015). History of artificial intelligence. Computer science, college of science, 1-6.
- [Result] Sönmez, D. (2009). Pediatrik yoğun bakım ünitesinde endotrakeal aspirasyon ağrısının değerlendirilmes, Yüksek lisans tezi, Marmara Üniversitesi Sağlık Bilimleri Enstitüsü, İstanbul.
- [Result] Terzi, B., Kaya, N. (2017). Konfor kuramı ve analizi. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 20: 1.
- [Result] Tutar Güven, Ş., & İşler Dalgıç, A. (2017). Prematüre yenidoğanlar için geliştirilmiş bireyselleştirilmiş destekleyici gelişimsel bakım programı. Uluslararası Hakemli Kadın Hastalıkları ve Anne Çocuk Sağlığı Dergisi, 9.
- [Result] Uga E, Candriella M, Perino A, Alloni V, Angilella G, Trada M, Ziliotto AM, Rossi MB, Tozzini D, Tripaldi C, Vaglio M, Grossi L, Allen M, Provera S. Heel lance in newborn during breastfeeding: an evaluation of analgesic effect of this procedure. Ital J Pediatr. 2008 Nov 18;34(1):3. doi: 10.1186/1824-7288-34-3. PMID 19490654
- [Result] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803
- [Result] Yıldırım, T. (2019). Sağlıkta dönüşüm ve yapay zekânın pediatriye yansımaları. Karadeniz Pediatri Günleri Kongre Özet Kitabı, 2 (1): 1-97.